CLINICAL TRIAL: NCT01046162
Title: An Open Label,Crossover,Randomized Study Of Two Periods,Two Treatments,Two Sequences, And A Single Dose Of Two Oral Drug Products Of Alprazolam 2mg (Tafil (r), Product Of Pharmacia& Upjohn S.a De C.v Vs Xanax 2mg, Product Of Pfizer Pharmaceuticals Llc) In Healthy Volunteers In Fasting Conditions
Brief Title: A Study Of Two Oral Preparations Of 2 Mg Alprazolam In Healthy Volunteers Under Fasting Conditions
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Collaborators: Investigacion Farmacologica y Biofarmaceutica, S.A. de C.V. (Other)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A6131021
Record Dates: First submitted 2010-01-07; First posted 2010-01-11 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Healthy
Keywords: Alprazolam; Tafil; Xanax; Bioequivalence; Drug Kinetics
MeSH Terms: interventions — Alprazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tafil Tablets 2 mg Pharmacia Upjohn (Active Comparator)
  Interventions: Drug: Alprazolam
- Xanax Tablets 2 mg Pfizer LLC (Active Comparator)
  Interventions: Drug: Alprazolam

INTERVENTIONS:
Drug: Alprazolam — Single tablet
  Other Names: Tafil Pharmacia Upjohn
  Arms: Tafil Tablets 2 mg Pharmacia Upjohn
Drug: Alprazolam — Single tablet
  Other Names: Xanax Pfizer
  Arms: Xanax Tablets 2 mg Pfizer LLC

SUMMARY:
The purpose of this study is to compare bioavailability between formulations of alprazolam in tablets to determine their bioequivalence in terms of rate and magnitude of absorption.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (male or female)
* Age between 18-40 years
* body mass index (Quetelet´s index) between 18-27

Exclusion Criteria:

* Unhealthy subjects
* Volunteers who require any medication over the course of the study
* Volunteers who have received investigational drugs within 60 days prior to the study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-07-15 (Actual); Primary Completion 2010-07-22 (Estimated); Study Completion 2010-07-22 (Estimated)

PRIMARY OUTCOMES:
Establish Cmax, Tmax, elimination half life, area below the curve from zero to t, and area below the curve from zero to infinity (ABC 0-∞) of the two formulations of Alprazolam. | 10 days
Statistically compare the bioavailability of the pharmaceutical formulations of Alprazolam studied, to establish or rule out the existence of bioequivalence. | 10 days

SECONDARY OUTCOMES:
Investigate the safety of both preparations based on the record of adverse events on completing both study periods. | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6131021&StudyName=A%20Study%20Of%20Two%20Oral%20Preparations%20Of%202%20Mg%20Alprazolam%20In%20Healthy%20Volunteers%20Under%20Fasting%20Conditions